CLINICAL TRIAL: NCT03518489
Title: Efficacy and Safety of Lappaconitine Adhesive Patch for the Treatment of Oral Mucositis Pain Caused by Chemoradiotherapy in Patients With Nasopharyngeal Cancer ： A Randomized, Prospective Single-center Controlled Study
Brief Title: Appaconitine Patch for Oral Mucositis Pain Caused by Chemoradiotherapy in Patients With Nasopharyngeal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FujianCH
Record Dates: First submitted 2018-04-23; First posted 2018-05-08 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Radiation Induced Oral Mucositis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Lappaconitine Adhesive Patch Lappaconitine Adhesive Patch is administered every radiation day, until the end of radiotherapy.
  Interventions: Drug: Lappaconitine Adhesive Patch
- Control (Active Comparator): Patients will be given standard care when oral pain is reported
  Interventions: Drug: standard care

INTERVENTIONS:
Drug: Lappaconitine Adhesive Patch — to evaluate the efficacy of lappaconitine adhesive patch in alleviation radiation induced mucositis pain
  Other Names: standard care
  Arms: Experimental
Drug: standard care — Standard care will include mouth wash with antibiotics.
  Arms: Control

SUMMARY:
The purpose of this clinical study is to evaluate the efficacy of lappaconitine adhesive patch in alleviation radiation induced mucositis pain and the improvements in QOL of patients with nasopharyngeal carcinoma . To determine if lappaconitine administered prior to radiation therapy reduces the severity of radiation induced oral mucositis pain in patients who have been diagnosed with nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a randomized, single -center study conducted in China to evaluate Lappaconitine Adhesive Patch in the reduction severity of radiation induced oral mucositis pain in patients receiving solo radiation therapy or chemoradiation therapy for nasopharyngeal carcinoma.

Patients will reveive daily fractions of IMRT (2.0 - 2.2 Gy) to a total of 60 - 72 Gy over approximately 7 weeks, plus cisplatin administered 80 - 100 mg/m2 once every three weeks for 3 doses or 30 - 40 mg/m2 once weekly for 6-7 doses (investigator's choice).

Patients in both arms received Intensity Modulated Radiation Therapy(IMRT) :All target volumes were outlined slice by slice on the axial contrast-enhanced CT with MR fusion images in the treatment planning system. The target volumes were defined in accordance with the International Commission on Radiation Units and Measurements Reports 50 and 62. The prescribed dose is 68-72 Gy to PTVnx (Planning target volume of the primary tumor), 64-68 Gy to GTVnd (Gross tumor volume of the cervical lymph node), 60- 64Gy to PTVnd and PTV1 (Planning target volume 1), and 54-58 Gy to PTV2 (Planning target volume 2) in 30-32 fractions.

Patients will be randomized equally to 1 of 2 treatment arms:

Arm A: Lappaconitine Adhesive Patch per day, concurrent with stardard care for oral mucositis Arm B: stardard care for oral mucositis

All patients will be assessed weekly for oral mucositis per WHO grading criteria until the completion of IMRT, and once weekly thereafter (if necessary) for 7 weeks, or until oral mucositis resolves to ≤ Grade 1.

Approximately 200 patients will be enrolled to ensure that roughly 80 patients per arm complete treatments for primary endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma without distant metastasis
* Clinical stage III~IVa( UICC (Union International Against Cancer) /AJCC (American Joint Committee on Cancer) TNM staging system 8th edition)
* Karnofsky Performance Status Scale between 60-100
* WBC count ≥ 4×109/L，neutrophil differential count≥ 1.5×109/L,Hemoglobin ≥ 90g/L， platelet count ≥ 100×109/L
* ALT or AST ≤2.5×ULN,bilirubin ≤2.5×ULN,Serum creatinine ≤1.5×ULN or Serum creatinine clearance≥60ml/min
* Sign the informed consent.

Exclusion Criteria:

* Younger than 18 years old or older than 70 years old
* Pregnancy or lactation
* Severe cerebrovascular disease/canker/psychosis/uncontrolled diabetes
* Have suffered from other tumor or now suffering from other tumor
* Have suffered from oral diseases or salivary gland diseases or mow suffering from oral diseases or salivary gland diseases
* Refuse to give up smoking/drinking/betel chewing
* suffering from other active infection diseases and in need of treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Numeric Rating Scale for Pain(NRS scale) at 7 weeks | The NRS scale will be assessed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks
  The pain caused by oral mucositis for all participants was assessed according to Numeric Rating Scale (NRS scale), by which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. And an 11-point scale where 0 indicates no pain and 10 indicates the worst imaginable pain. The scale for each patient was recorded.

SECONDARY OUTCOMES:
Incidence of Severe Acute Oral Mucositis (Grade of CTCAE ≥ 2) | The WHO score will be assessed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks.
  The Oral Mucositis Score of World Health Organization (WHO) was classified based on the changes of patients' oral mucosa and ability to eat, and are classified to 4 grades. WHO scale for oral mucositis (available in: Peterson DE, Boersdoets CB, Bensadoun RJ, et al. Management of oral and gastrointestinal mucosal injury: ESMO Clinical Practice Guidelines for diagnosis, treatment, and follow-up. Annals of Oncology 2015; 26(supply5). https://doi.org/10.1093/annonc/mdv202 ): Grade 0 = no oral mucositis; Grade 1 = erythema and soreness; Grade 2 = ulcers, able to eat solids; Grade 3 = ulcers, requires liquid diet (due to mucositis); Grade 4 = ulcers, alimentation not possible (due to mucositis).
Change from Baseline Quality of Life at 7 weeks | The EORTC QLQ-C30 shoule be completed weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks.
  he quality of life for all participants was evaluated according to The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) (available in: Grønvold M. EORTC QLQ-C30 Scoring Manual 2014.)
Change from Baseline Karnofsky Performance Status Scale at 7 weeks | The KPS Scale will be recoreded weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks
  The functional status for all participants was assessed according to Karnofsky Performance Status Scale (KPS Scale) (available in: Friendlander AH, Ettinger RL. Karnofsky performance status scale[J]. Special Care in Dentistry, 2009, 29(4):147.). The KPS Scale was range from 0 to 100, and were averagely divided into eleven grades begin with 0.
The Adverse events Related to lappaconitine | The Adverse events Related to lappaconitinewill be recoreded weekly during concurrent chemoradiotherapy (CCRT) for 7 weeks.
  The adverse events related to lappaconitine based on medicine specification of lappaconitine was observed and recorded down according to Common toxicity criteria, version 2.0. (available in: Version CTC, Version CTC, Date P, et al. Common toxicity criteria (ctc) 1999.)

CONTACTS AND LOCATIONS:
Overall Officials: Shufang Qiu, M.D., Study Director — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer Hospital Radiation Oncology Department, Fuzhou, Fujian, China